CLINICAL TRIAL: NCT01489774
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Single/Multiple Dose, Dose-escalation Clinical Study to Investigate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of CJ-12406 After Oral Administration in Healthy Male Subjects, Phase I Study
Brief Title: Phase I Study to Investigate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of CJ-12406 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CJ_HET_101
Record Dates: First submitted 2011-11-09; First posted 2011-12-12 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Digestive System Diseases
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CJ-12406 (Experimental): CJ-12406 Tablet, daily for 1 day or bid for 10 days
  Interventions: Drug: CJ-12406

INTERVENTIONS:
Drug: Placebo — single and multiple dose
  Arms: Placebo
Drug: CJ-12406 — single and multiple dose
  Arms: CJ-12406

SUMMARY:
Study objectives

* To evaluate the safety, tolerability, and pharmacokinetics of escalating single oral doses of CJ-12406 in healthy male subjects.
* To evaluate the pharmacodynamics of CJ-12406 after multiple oral administrations to healthy male subjects.
* To evaluate the effect of food on the pharmacokinetic of a single oral dose of CJ-12406 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male volunteers in the age between 20 and 45 years old
2. Subjects with no history of any significant chronic disease
3. The weight range is not exceed ±20% of ideal weight. Ideal weight = [height -100]*0.9
4. Judged to be in good health on the basis of their vital sign, ECG, physical exam and routine laboratory data
5. Available for the entire study period
6. Willing to adhere to protocol requirements and sign a informed consent form
7. Multiple escalation study; H. pylori positive, as determined by the urea breath test

Exclusion Criteria:

1. History of clinically significant allergies including drug allergies
2. History of clinically significant hepatic, renal, gastrointestinal, pulmonary, ,musculoskeletal, endocrine, psychiatric, hematologic, oncologic, neurologic or cardiovascular disease
3. Symptom of an acute illness within 4 weeks prior to drug administration
4. History of surgery except or gastrointestinal diseases which might significantly change absorption of medicines
5. Treatments or symptoms of symptomatic GERD, gastric ulcer, duodenal ulcer, functional dyspepsia, irritable bowel syndrome within 3 months prior to drug administration
6. Clinical laboratory test values are outside the accepted normal range

   * AST or ALT >1.25 times to normal range
   * Creatinine clearance <80 mL/min
   * 12-lead ECG; PR ≥ 210 msec, QRS ≥ 120 msec, QT ≥ 500 msec, QTcF ≥ 450 msec
7. Clinically significant vital signs

   * Hypotension (SBP ≤ 89 mmHg)
   * Hypertension (SBP ≥ 141 mmHg or DBP ≥ 91 mmHg)
   * Tachycardia (≥ 101 beats/min)
8. History of drug and alcohol abuse(alcohol > 30 g/day)
9. Subjects who have ever smoke within 3 months prior to drug administration
10. Positive urine screen for drugs and cotinine
11. Use of any other medication, including herbal products, within the 2 weeks before dosing
12. Special diet known to interfere with the absorption, distribution, metabolism or excretion of drugs (especially, consumption of grapefruit juice) within 7 days prior to drug administration
13. Donated blood within 60 days prior to dosing
14. Participated in a previous clinical trial within 90 days prior to dosing
15. Subjects considered as unsuitable based on medical judgement by investigators

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of CJ-12406 | 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose
  Blood samples were collected before dosing and 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose (multiple dose study; 1 and 10 day). For multiple dose study, additional blood samples will be drawn predose (immediately prior to morning dosing) on days 3, 7, and 9.
Number of participants with adverse events | A range of 17 days - from screening to gollow-up visit
Peak plasma concentration (Cmax) of CJ-12406 | 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose
  Blood samples were collected before dosing and 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose (multiple dose study; 1 and 10 day). For multiple dose study, additional blood samples will be drawn predose (immediately prior to morning dosing) on days 3, 7, and 9.
Area under the plasma concentration versus time curve (AUC) of active metabolite | 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose
  Blood samples were collected before dosing and 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose (multiple dose study; 1 and 10 day). For multiple dose study, additional blood samples will be drawn predose (immediately prior to morning dosing) on days 3, 7, and 9.
Peak plasma concentration (Cmax) of active metabolite | 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose
  Blood samples were collected before dosing and 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post dose (multiple dose study; 1 and 10 day). For multiple dose study, additional blood samples will be drawn predose (immediately prior to morning dosing) on days 3, 7, and 9.

SECONDARY OUTCOMES:
H. pylori eradication rate | 38 days post dose (plus of minus 1 day)
  UBT test
The percent time of intragastric pH>4 | 7 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, MD. PhD, Principal Investigator — Inje University
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea